CLINICAL TRIAL: NCT06670183
Title: The Associations Between Diet and Rheumatoid Arthritis Risk in the UK Biobank
Brief Title: Dietary Factors and Rheumatoid Arthritis Risk in the UK Biobank
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Darren Greenwood, Senior Lecturer in Biostatistics, University of Leeds
Other Study IDs: fsydo_UKBB
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Nutrition; Rheumatoid Arthritis; Body Mass Index; Alcohol consumption; Cohort study; Epidemiology; Arthritis, Rheumatoid, Seropostive
MeSH Terms: conditions — Arthritis, Rheumatoid; Alcohol Drinking; Arthritis | interventions — Dietary Patterns; Nutrients; Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — UK Biobank collected biomarker samples with DNA. This project makes use of data from the biomarker samples, but no additional samples will be taken and no additional samples will taken for this research. No samples will be processed, stored or retained by us. For the previously published details of UK Biobank, with anonymised data made available for researchers, please see: https://www.ukbiobank.ac.uk/enable-your-research/about-our-data/biomarker data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- UK Biobank: UK Biobank. There are no interventions in this observational cohort study.
  Interventions: Other: Dietary patterns; Other: Food groups and Nutrients; Other: Alcohol intake; Other: Vitamin D status

INTERVENTIONS:
Other: Dietary patterns — Dietary patterns such as regular meat-eater, occasional meat-eater, pescatarian, and vegetarian; Mediterranean diet.
Other: Food groups and Nutrients — Dietary components, such as oily fish, dairy product, supplements, fibre, vitamin D supplements.
Other: Alcohol intake — Frequency and intake of alcoholic beverages was measured by self-reporting the weekly frequency of different types of alcoholic beverages, e.g., the number of pints of beer/cider consumed per week and measures of spirits or liquors consumed per week were collected to assess consumption of beer/cider and spirits.
Other: Vitamin D status — Serum 25(OH)D was measured once at baseline through a non-fasted blood draw during any season of the year.

SUMMARY:
Rheumatoid arthritis (RA) is the most common inflammatory arthritis, affecting around 1% of the UK population. It affects around 400,000 adults and is characterised by synovial inflammation, cartilage and bone damage that requires lifelong treatment and represents a significant burden for both the individual and society. Diet can affect inflammatory status and RA risk, with varying risks for men and women on specific diets. People with low to moderate consumption of alcohol may be at a lower risk of RA. Those who consume lower intakes of fruit and vegetables could be at a greater risk than those with adequate intakes. This research aims to better understand the role of diet in reducing RA risk in men and women in the United Kingdom. The research will use existing dietary and lifestyle data from the United Kingdom Biobank Study and hospital records of RA incidence.

DETAILED DESCRIPTION:
Background:

RA is the most common inflammatory arthritis in the United Kingdom, contributing significantly to increased morbidity and mortality, particularly from cardiovascular diseases. Epidemiological evidence suggests that compared to occasional drinkers, moderate alcohol consumption may reduce RA risk compared to non-drinkers, and occasional drinking. Additionally, observational research highlights the potential for RA risk reduction through dietary modifications, though evidence on interactions between dietary and genetic factors remains limited, particularly in prospective cohort studies. Moreover, the mechanisms underlying potential differences in RA risk between men and women are not yet fully understood.

This study aims to assess the associations between dietary factors, such as alcohol consumption and dietary patterns, and RA incidence within the UK Biobank cohort. A secondary objective is to evaluate the role of potential modifiers in the relationship between dietary factors and RA risk, including adherence to the Alternative Healthy Eating Index (AHEI), Townsend index, as well as age, sex, body mass index (BMI), smoking status, and physical activity. Additionally, interactions between dietary factors and genetic profiles in relation to RA risk will be investigated.

Research plan and methods:

This study will utilize dietary and lifestyle data from the UK Biobank, a cohort that recruited over 500,000 adults from 2006 to 2010, and linked hospital records to identify incident RA cases.

Cox proportional hazards regression models will be employed to examine associations between dietary factors and RA incidence, adjusting for relevant confounders. Potential effect modifiers such as age, sex, AHEI score, Townsend index, BMI, smoking status, physical activity, and gene-diet interactions will be analyzed by including interaction terms in the Cox models. Causal mediation analysis will further clarify the role of potential mediators. Additionally, inflammatory and immune-related factors, metabolic profile, and genetic susceptibility will be assessed to explore their contributions to RA risk.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Ages 40 to 70 years at time of recruitment
* Able to provide informed consent

Exclusion Criteria:

* Unable to link dietary and lifestyle data with hospital episode statistics
* Had a rheumatoid arthritis before or no the date of recruitment
* Withdrew consent during the study period
* Genetic sex differs to reported sex
* Outlier diet or anthropometric data (energy intake <500 or >5000 kcal/day or body mass index <10 or >60 kg/m2)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population. Information on the UK Biobank cohort profile is available here: https://www.ukbiobank.ac.uk/
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Rheumatoid Arthritis incidence (first) | Time Frame: Age when the completed questionnaire was returned (2006-2010) until age at event, death, or end of study period (2024).
  First RA incidence, identified from all relevant ICD diagnosis codes and treatment codes identified through linked HES data.

CONTACTS AND LOCATIONS:
Overall Officials: Darren C Greenwood, PhD, Principal Investigator — University of Leeds

IPD SHARING:
Plan to Share IPD: Yes
IPD from UK Biobank is available to genuine researchers on application (https://www.ukbiobank.ac.uk/enable-your-research/apply-for-access).
Supporting Information: Study Protocol, ICF
Time Frame: IPD from UK Biobank is available to genuine researchers on application (https://www.ukbiobank.ac.uk/enable-your-research/apply-for-access).
Access Criteria: IPD from UK Biobank is available to genuine researchers on application (https://www.ukbiobank.ac.uk/enable-your-research/apply-for-access).
URL: https://www.ukbiobank.ac.uk/enable-your-research/apply-for-access

REFERENCES:
- [Background] Sudlow C, Gallacher J, Allen N, Beral V, Burton P, Danesh J, Downey P, Elliott P, Green J, Landray M, Liu B, Matthews P, Ong G, Pell J, Silman A, Young A, Sprosen T, Peakman T, Collins R. UK biobank: an open access resource for identifying the causes of a wide range of complex diseases of middle and old age. PLoS Med. 2015 Mar 31;12(3):e1001779. doi: 10.1371/journal.pmed.1001779. eCollection 2015 Mar. PMID 25826379
- See also: Study website — https://www.ukbiobank.ac.uk/